CLINICAL TRIAL: NCT05490758
Title: Comparison of Sensorimotor Training and Constraint Induced Movement Therapy on Upper Extremity Function in Children With Hemiplegic Cerebral Palsy
Brief Title: Sensorimotor Training and Constraint Induced Movement Therapy on Upper Extremity Function in Children With Hemiplegic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0718
Record Dates: First submitted 2022-07-14; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: sensorimotor training; motor function; constraint induced movement therapy
MeSH Terms: interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensorimotor training (Experimental): sensorimotor training group did sensorimotor activities e.g play with dough,peg games 5 days a week for 4 weeks.
  Interventions: Other: sensorimotor training
- constraint induced movement therapy (Experimental): constraint induced movement therapy group in which affected arm was constraint for 6 hours a day for 5 days a week for 4 weeks.
  Interventions: Other: constraint induced movement therapy

INTERVENTIONS:
Other: sensorimotor training — sensorimotor training include activities like play with dough, peg games, puzzles for 5 days a week for 4 week.
  Arms: sensorimotor training
Other: constraint induced movement therapy — constraint induced movement therapy in which arm was constraint for 6 hours a day for 5 days a week for 4 week.
  Arms: constraint induced movement therapy

SUMMARY:
The aim of the work was to find out the effects of sensorimotor training and constraint induced movement therapy on upper extremity function in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
The significance of this study is that there was paucity of literature in finding the comparative effects of sensorimotor training and constraint induced movement therapy on upper extremity function in children with hemiplegic cerebral palsy. The aim is to find out the effects of sensorimotor training on motor functioning of the upper extremity in comparison of constraint induced movement therapy.

ELIGIBILITY:
Inclusion Criteria:

* subjects who were fully oriented
* children diagnosed with hemiplegic cerebral palsy
* no history of intramuscular botulinum injections past one year

Exclusion Criteria:

* children with epilepsy
* gross deformity of upper limb
* children with contractures

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
nine hole peg test | 4 weeks
  nine hole peg test to check hand dexterity and grip. The patient is seated at a table with a container holding nine pegs and a wood/plastic block containing nine empty holes and asked to put the nine pegs in nine holes in a block one by one and then remove the pegs one at a time from the holes and the time is recorded. patient should do the test with both hands independently.

SECONDARY OUTCOMES:
manual ability classification system | 4 weeks
  it describes how CP child uses his or her hands to handle objects in daily activities with qualitative analysis by care taker, it has five levels. in level 1 child holds objects easily and succesfully. in level 2 child handles most object but with some reduced quality or speed. in level 3 the objects are handled with difficulty and child needs help to prepare or modify activities. in level 4 child handles a limited selection of easily managed objects and always requires some help from others. in level 5 child is not able to handle objects or to complete even simple actions with their hands.

OTHER OUTCOMES:
two point discrimination | 4 weeks
  two point discrimination to discern that the two nearby objects touching the skin are truly two distant points. it is tested with a sharp object caliper is applied to the exposed skin and response and time are recorded. it is used for tactile perception. the normal minimal distance for the hands is 3cm and 0.6 cm for the fingers tips.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, PhD, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoare BJ, Wallen MA, Thorley MN, Jackman ML, Carey LM, Imms C. Constraint-induced movement therapy in children with unilateral cerebral palsy. Cochrane Database Syst Rev. 2019 Apr 1;4(4):CD004149. doi: 10.1002/14651858.CD004149.pub3. PMID 30932166
- [Background] Santana CAS, Tudella E, Rocha NACF, de Campos AC. Lower Limb Sensorimotor Training (LoSenseT) for Children and Adolescents with Cerebral Palsy: A Brief Report of a Feasibility Randomized Protocol. Dev Neurorehabil. 2021 May;24(4):276-286. doi: 10.1080/17518423.2020.1858458. Epub 2021 Jan 3. PMID 33393402
- [Background] Samaei A, Mirshoja MS, Khalili MA. Comparison of Sensorimotor Retraining Methods by Movement Therapy Based on Limitations in Upper Extremity Function in Patients with Chronic Stroke. INTERNATIONAL JOURNAL OF PHARMACEUTICAL RESEARCH AND ALLIED SCIENCES. 2016;5(2):510-+.